CLINICAL TRIAL: NCT06320860
Title: FlexStone Enabled Kidney Stone Retrieval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoTheia (Industry)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB231189
Record Dates: First submitted 2024-03-08; First posted 2024-03-20 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Kidney Stone Retrieval (Experimental): All patients in this group will have the EndoTheia FlexStone basket used to assist in the retrieval of kidney stones
  Interventions: Device: Kidney Stone Retrieval

INTERVENTIONS:
Device: Kidney Stone Retrieval — Using FlexStone Basket aimability to retrieve kidney stones

SUMMARY:
This study investigates if additional basket control in helpful during retrieval of kidney stones especially those that are difficult to reach for standard baskets.

DETAILED DESCRIPTION:
The clinical practice at Vanderbilt University Medical Center will perform standard flexible ureteroscopy (fURS) procedures using conventional stone retrieval baskets, the EndoTheia FlexStone basket, laser fibers for intracorporeal lithotripsy , and any other fURS accessory devices as determined by the surgeon. If renal calculi are present which the physician deems retrieval of would benefit from the added aimability of the EndoTheia FlexStone basket will be used.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 80 years of age
* Able to provide written informed consent
* Have renal stones present and are appropriate candidates for fURS

Exclusion Criteria:

* Females who are pregnant. As part of routine pre-operative care, all females of childbearing potential will undergo either urine or blood pregnancy testing.
* Cancer positive subjects or any patients currently undergoing any treatment or therapy to treat, cure, or mitigate cancer.
* Patients with active urinary tract infection or anatomy that complicates retrograde access to the ureter and kidney
* Patients who do not meet inclusion criteria
* Patients who are unable or unwilling to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Successful retrieval of kidney stones | Day 1 Post-Intervention
  The primary end point of this feasibility study is to demonstrate that the additional basket aimability of the device enables basket to capture stones in difficult to reach locations such as the lower pole.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States